CLINICAL TRIAL: NCT02660775
Title: Social Cognitive Assessment in Psychiatry - Validation of a New Battery: ClaCoS
Brief Title: Social Cognitive Assessment in Autism and Schizophrenia
Acronym: (ClaCoS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-A00580-49
Record Dates: First submitted 2015-12-16; First posted 2016-01-21 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- schizophrenia (Experimental): this project is to assess relevance of ClaCoS in schizophrenia compared to healthy controls, and to analyze links between social cognition and both neurocognition and symptoms, (2) to collect data in a large sample of healthy controls in order to establish appropriate standards for tools composing ClaCoS battery.
  Interventions: Behavioral: schizophrenia
- autism (Experimental): this project is to assess relevance of ClaCoS in autism compared to healthy controls, and to analyze links between social cognition and both neurocognition and symptoms, (2) to collect data in a large sample of healthy controls in order to establish appropriate standards for tools composing ClaCoS battery.
  Interventions: Behavioral: Autism
- healthy controls (Placebo Comparator): this project is to assess relevance of ClaCoS in autism compared to healthy controls, and to analyze links between social cognition and both neurocognition and symptoms, (2) to collect data in a large sample of healthy controls in order to establish appropriate standards for tools composing ClaCoS battery.
  Interventions: Behavioral: Healthy controls

INTERVENTIONS:
Behavioral: schizophrenia — The battery (ClaCoS) is composed by 6 tests and several scores will be recorded for each:
  * for emotion perception : Facial emotions recognition task (TREF)
  * for theory of mind : Movie for the assessment of social cognition ( MASC-VF)
  * for attributional bias : Ambiguous Intentions Hostility Questionnaire ( AIHQ)
  * for social perception and knowledge : interpretation score - with and without index, comprehension score ( PerSo )
  * for empathy :Questionnaire of cognitive and affective empathy ( QCAE) for people with schizophrenia
  * for self assessment : Self - assessment of social cognition (ACSo)
  Arms: schizophrenia
Behavioral: Autism — The battery (ClaCoS ) is composed by 6 tests and several scores will be recorded for each:
  * for emotion perception : Facial emotions recognition task(TREF ): total score, score per emotion, detection levels
  * for theory of mind : Movie for the assessment of social cognition (MASC ) :total score, error type
  * for attributional bias : Ambiguous Intentions Hostility Questionnaire (AIHQ) :hostility score, attribution score, aggression score
  * for social perception and knowledge : interpretation score - with and without index, comprehension score ( PerSo )
  * for empathy : Empathy quotient (EQ)
  * for self assessment : Self - assessment of social cognition ( ACSo ): total score and scores per processes
  Arms: autism
Behavioral: Healthy controls — only social cognitive measures
  Arms: healthy controls

SUMMARY:
In people with schizophrenia or people with autism, impairments of social cognition are a core feature of the disease and, according to researchers who represent valuable references on this subject for the international community, three to five processes of social cognition are usually altered in those diseases: (1) emotional processing which is the ability to identify emotions through facial expressions, gestures, and tone of voice, (2) theory of mind (ToM), which is defined as "the ability to attribute mental states (beliefs, intents, desires, …) to oneself and others, and to understand that others have beliefs, intentions, and desires that are different from one's own", (3) attributional style which refers to how people explain the causes of positive and negative events, and corresponding, in schizophrenia, to self-serving and personalizing bias that means a tendency to blame others for negative life events rather than sharing the responsibilities between different sources; and (4 and 5) social perception and knowledge, which can be defined as decoding and interpreting social cues from others, taking the social context into account, and knowing social rules, roles, and goals. Components of social cognition appear to be related to both symptomatology and functioning in everyday life. The present study aims to assess a new social cognitive battery developed by several teams in France: ClaCoS.

DETAILED DESCRIPTION:
The project's objectives are: (1) to assess relevance of ClaCoS in schizophrenia and autism compared to healthy controls, and to analyze links between social cognition and both neurocognition and symptoms, (2) to collect data in a large sample of healthy controls in order to establish appropriate standards for tools composing ClaCoS battery.

For the first objective, three kind of evaluation will be proposed: clinical, neurocognitive and social cognitive (ClaCoS). Three populations of 80 participants will be compared: healthy controls, patients with schizophrenia or schizoaffective disorders, and patients with autism spectrum disorders. These three groups will be matched on sex, age and level of education.

For the second objective a systematic collection of data will be carried out in a large sample of healthy controls. In this part of the study, only social cognitive measures will be recorded. Subjects will be ranked according to three criteria: three classes for age (18-25 years old, 26-35 and 36-45), five classes for socio-professional status according to the INSEE classification, and two classes for sex (men/women).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years old
* No psychiatric or neurologic conditions or comorbidity
* No relatives with people with people with history of neuropsychiatric disease
* French native language or education in a French school since the first year of primary school
* Consent to participate to the study

Exclusion Criteria:

* Aged 18-45 years old
* Patients with schizophrenia: diagnosis assessed with DSM5 criteria
* No modification of psychotropic treatment during the month before inclusion
* French native language or education in a French school since the first year of primary school
* Consent to participate to the study and agreement of the legal guardian

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in social cognition measures | Week 12
  The battery (ClaCoS ) is composed by 6 tests and several scores will be recorded for each:
  * for emotion perception : total score, score per emotion, detection levels (TREF)
  * for theory of mind : total score, error type (MASC)
  * for attributional bias : hostility score, attribution score, aggression score (AIHQ )
  * for social perception and knowledge : interpretation score - with and without index, comprehension score (PerSo)
  * for empathy : Empathy quotient (EQ) for people with autism / Questionnaire of cognitive and affective empathy (QCAE )for people with schizophrenia (total score and sub scores)
  * for self assessment : total score and scores per processes( ACSo )

SECONDARY OUTCOMES:
Change from Baseline in symptoms measure | Week 12
  Positive and negative symptoms scale, global score, positive sub scale score and negative sub scale score (PANSS)
Change from Baseline in Neurocognitive functioning measures | Week 12
  Several neurocognitive processes will be assessed and notably memory, attention, executive functions, and processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK NICOLAS, PUPH, Principal Investigator — Service Universitaire de Réhabilitation - Le Vinatier Hospital
Locations (1):
- Professeur FRANCK Nicolas, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No